CLINICAL TRIAL: NCT00843648
Title: Study of the Development of Human Immune System of Newborns by Antigen Chips
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Center
Other Study IDs: SHEBA-08-5441-AM-CTIL
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Antibody Immune Profile
Keywords: antibody immune profile; preterm; c-section; breastfeeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- preterms: mother and preterm babies
- term-bfing: term breastfed babies and mothers
- term-PIF: term non breastfed babies and mothers
- c-section: c-section babies and their mothers

SUMMARY:
The immune system is a dynamic, constantly evolving network. Excluding autoimmune diseases, healthy individuals are also known to have a large number of circulating antibodies that can recognize proteins of their own tissues. These antibodies are known as natural antibodies and previous studies suggested that some features of these "self" components are shared by individuals in certain physiological states. Thus, monitoring self immunoglobulins can provide an overview of the various states of the immune system. To do so, and in the process to obtain systems biology view of the immune system, the newly developed Antigen Chip technology has been used.

To further investigate this subject we plan to carry out broader investigations that will be conducted in collaboration with the group of Prof. Eshel Ben-Jacob from the university of Tel-Aviv and Prof. Irun Cohen from the Weizmann Institute that have the required experimental and analytical expertise and facilities. The studies will include follow-up on the immune state of babies and their mothers for several months post birth using the Antigen Chip and analyzed by the Immune holography method. The investigations will also include comparative studies between the immune signature of different body fluids, the effects of feeding, and the effect method and time of labor.

DETAILED DESCRIPTION:
Antibody reactivities are traditionally studied by their individual reactivities to one or only a few antigens, whereas only a small number of studies have focused on the repertoires of antibodies to large numbers of defined antigens. Only recently, a new technology for system level analysis, the immune microarrays (or antigen chips) was introduced [Quintana 2004, Quintana and Cohen 2004, Robinson 2006]. This technology is capable of detecting patterns of antibodies binding to many hundreds of antigens, foreign or self and thus allowing a systems biology view of immune system. To create the antigen chips, a robotic apparatus is used to spot the antigen molecules of choice - proteins, peptides, sugars, lipids, nucleic acids - to a coated glass slide. These antigens are covalently linked to the surface of the slide and a drop of blood serum or any other body fluid can be tested for antibodies binding to hundreds of these antigen spots. The subject's bound antibodies are detected using fluorescence-labeled second antibodies and the reactions are monitored by laser activation.

ELIGIBILITY:
Inclusion Criteria:

* Term and preterm newborns and their mothers
* Age 1 day to 7 weeks

Exclusion Criteria:

* Maternal immune dieases
* Major congential malformations

Ages: 1 Day to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: term and preterm newborns and their mothers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel